CLINICAL TRIAL: NCT05329688
Title: The Effect of Nutrition Education Program on the Nutrition Status and Life Quality of Cancer Patients Receiving Radiotherapy
Brief Title: Nutrition Education Program for Cancer Patients Receiving Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Asia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB110-196-A
Record Dates: First submitted 2022-04-07; First posted 2022-04-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-04

CONDITIONS: Radiotherapy Side Effect; Nutrition Related Cancer
Keywords: nutrition; radiotherapy; cancer patients
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Intervention Model Description: single blind (Participant)
Who Masked: Participant
Masking Description: single blind (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Novel nutrition program :
  Give nutrition health education every week and regular survey and intervention. The education booklets are made based on the guideline and characteristics of the disease.
  Interventions: Procedure: novel nutrition program
- Arm B (Active Comparator): Routine nutrition education Give nutrition education if the patient visits the clinics. Irregular survey and intervention were given to the patients.
  Interventions: Procedure: novel nutrition program

INTERVENTIONS:
Procedure: novel nutrition program — Give nutrition health education every two weeks and regular survey and intervention. The education booklets are made based on the guideline and characteristics of the disease.

SUMMARY:
Using randomized control study, explore the effect of novel nutrition education program on the nutrition status and life quality of cancer patients receiving radiotherapy

DETAILED DESCRIPTION:
Weight loss is common among cancer patients, and can be attributed to many causes, including mucositis, inability to ingest or absorb adequate calories because of a problem with the alimentary tract, loss of appetite, and metabolic aberrations. Unintentional weight loss may be associated with decreased quality of life (QOL) and a poorer prognosis. Furthermore, for patients who are already in a catabolic state, the increased metabolic demands associated with anticancer treatment (particularly surgery) further worsen the problem. The novel nutrition program might improve the nutrition status and QOL in cancer patients receiving radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are diagnosed with cancer and receive radiotherapy, especially in head and neck cancer, lung cancer, or esophageal cancer.
2. Patients need nutrition support treatment
3. Informed consent

Exclusion Criteria:

1. Critical patients or life expectancy < 12 weeks
2. Patients with severe hepatic cirrhosis, Chronic Obstructive Pulmonary Disease, chronic renal failure, intestinal obstruction, stroke.
3. Unconscious or psychiatric patients
4. Patients with communication problems

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
risk of malnutrition | Week 0, 12
  Nutrition Risk Screening 2002 is used to assess the risk of malnutrition.
BMI | Week 0, 12
  Body mass index is a measure of body fat based on height and weight that applies to adult men and women. It equals to weight divided by height square.
albumin | Week 0, 12
  level of serum albumin
Quality of Life (QOL) | Week 0, 12
  The QOL was measured by the European Organization for Research and Treatment quality of life version 3 questionnaire (EORTC QLQ-C30) simplified Chinese version. It contains five functional scales (physical, role, cognitive, emotional, and social), three symptoms scales (fatigue, pain, and nausea and vomiting), a global health scale, a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnea, appetite loss, insomnia, constipation, and diarrhea) and financial impact of the disease. For most items, four response categories from 1 (not at all) to 4 (very much) are employed; two items (overall health, overall quality of life) have response categories ranging from 1 to 7. A high scale score represents a higher response level. Thus a high score for a functional scale, the global health status or overall QOL represents a high or healthy status or a high QOL; however, a high score for the symptom scales represents a high level of symptom.

SECONDARY OUTCOMES:
physical function status | Week 0, 12
  Using Eastern Cooperative Oncology Group to assess the physical function.
Knowledge-Attitude-Practice | Week 0, 12
  Knowledge Scale composes of 10 questions and 10 scores for each question. Attitude and Practice Scale have 5 questions. Each question is rated as A、B、C. A represents 20 score and B is 10 score.

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Yuan Wu, Study Director — Asia University, Taiwan
Locations (1):
- Szu-Yuan Wu, Taipei, Please Select, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
study completed
Supporting Information: Study Protocol
Time Frame: data will become available on June 30 2022.
Access Criteria: requirement with official application